CLINICAL TRIAL: NCT02982278
Title: Wide Spectrum Investigation of Stroke Outcome Disparities on Multiple Levels (WISSDOM): Community-based Intervention Under Nurse Guidance
Brief Title: Wide Spectrum Investigation of Stroke Outcome Disparities on Multiple Levels (WISSDOM)
Acronym: CINGS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: PRO 46339
Record Dates: First submitted 2016-12-01; First posted 2016-12-05 (Estimated); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Stroke Ischemic; Minority Health
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CINGS Intervention (Experimental): CINGS is a 12-week nurse coordinated, Community Health Worker (CHW) intervention structure. Registered Nurse (RN) developed After hospital care plan with home visits sessions will be conducted by the CHW and intermittent televideo RN interactions. After baseline assessment, participants randomized to the intervention group will have home visits, once a week for the first month, and biweekly during months two and three. follow up assessments at 3, 6, and 12-month intervals.
  Interventions: Behavioral: Community-based Intervention under Nurse Guidance after Stroke
- Control (Experimental): Control group will receive usual care. Base line visit and follow up at 3, 6, and 12 months post stroke enrollment.
  Interventions: Behavioral: Community-based Intervention under Nurse Guidance after Stroke

INTERVENTIONS:
Behavioral: Community-based Intervention under Nurse Guidance after Stroke — CINGS is a 12-week nurse coordinated, Community Health Worker intervention structure. Intervention home visits will be conducted by the CHW and will include home-based training in self-care and self-management strategies alongside strategies to address risk of negative stroke outcomes that will be determined once these risk factors are identified and community-engaged approaches to their resolution derived. CHW efforts will be guided via televideo interactions with nurse coordinator. During home-visits, self-reported assessments will be collected via RedCap as well as assessments collected by the CHW and research nurse (weight, blood pressure, medication adherence). After baseline, participants randomized to the intervention group will have home visits, once a week for the first month, and biweekly for the other two months, conducted by the CHW. Additionally, there will be post-intervention follow-up assessments at 3, 6, and 12-month time intervals.
  Other Names: CINGS

SUMMARY:
This research project will evaluate the relationship between cardiovascular risk factors, degrees of physical and mental activity prior to the stroke, brain tissue integrity, post-stroke community participation and neurological recovery after the stroke. Investigators will recruit and study healthy and post stroke participants, gaining insight into the possible mechanisms that explain why the adverse risk profile, which is more commonly present in African-Americans than non-Hispanic Whites in the stroke belt, is translated into a less favorable recovery post stroke.

DETAILED DESCRIPTION:
Stroke is a common cause of disability, but not all subjects who survive a stroke are left with debilitating sequelae. The human brain is able to self-repair and adapt after injury through neuroplasticity, which is crucial for stroke recovery. At present, recovery cannot be completely predicted from clinical stroke variables. A promising theory suggests that the health status of the stroke host is as important as stroke severity for recovery. Within the neurological system, health is reflected by the integrity of the brain tissue and its neuronal environment, which provide the neuroplastic potential that is necessary for recovery. The potential for neuroplasticity is likely variable across individuals and possibly accounts for some of the differences in outcome that cannot be explained by other clinical factors.

A better understanding of the relationship between stroke outcomes, host brain tissue integrity and recovery environment would have immense potential to address stroke related disabilities. The investigators are experts in research involving brain tissue integrity using neuroimaging and recovery environment using community based participation approaches involving nurse-guided community health workers (CHWs).

This research project will evaluate the relationship between cardiovascular risk factors, degrees of physical and mental activity prior to the stroke, brain tissue integrity, post-stroke community participation and neurological recovery after the stroke. The investigators will recruit and study a biracial cohort, gaining insight into the possible mechanisms that explain why the adverse risk profile, which is more commonly present in African-Americans than non-Hispanic Whites in the stroke belt, is translated into a less favorable recovery post stroke. If a better understanding of the underlying reasons for this observation can be defined, an important first step toward eliminating this disparity can be achieved.

ELIGIBILITY:
Inclusion Criteria:

* 40-75 years
* prestroke mRS score >2
* African American or White
* Reside in Berkeley, Charleston, Dorchester, Colleton or Georgetown Counties
* Ischemic stroke involving only one hemisphere
* Fugl Meyer score >16 at baseline or Aphasia Quotient in Western Aphasia Battery <93
* no contraindications to research MRI

Exclusion Criteria:

* Primary or secondary intracerebral hematoma, or subarachnoid hemorrhage, or subdural/ epidural hematoma; Prisoner; diagnoses of substance addiction (alcohol or illicit drugs)
* Bihemispheric acute ischemic strokes;
* Other concomitant neurological disorders, such as brain tumor, abscess or spinal cord disease affecting language or limb motor function;
* Documented history of dementia prior to index event;
* Patient suffered one or more recurrent stroke during the 12-month follow up period.
* Terminal illness with life expectancy ≤ 1 year
* Currently pregnant
* Brain stem strokes

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Stroke Specific Quality of Life Scale | 3, 6, 12 months
  Quality of Life
Stroke Impact Scale | 3, 6, 12 months
  Stroke recovery
NIH Stroke Scale | 0, 3, months
  Stroke Severity

SECONDARY OUTCOMES:
Medical Outcomes Study Social Support Scale | 3, 6, 12 months
  Social Support
Patient Health Questionnaire-9 | 3, 6 12 months
  Depression

OTHER OUTCOMES:
Stroke Self-Efficacy Scale | 3, 6, 12
  Self-efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Gayenell Magwood, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Buie JNJ, Zhao Y, Burns S, Magwood G, Adams R, Sims-Robinson C, Lackland DT; WISSDOM Research Center Study Group. Racial Disparities in Stroke Recovery Persistence in the Post-Acute Stroke Recovery Phase: Evidence from the Health and Retirement Study. Ethn Dis. 2020 Apr 23;30(2):339-348. doi: 10.18865/ed.30.2.339. eCollection 2020 Spring. PMID 32346280